CLINICAL TRIAL: NCT07116681
Title: The Acute Effects of Dry Powder Inhaled Treprostinil on Stroke Volume Augmentation and Dead Space Ventilation in Patients With Exercise-induced Pulmonary Hypertension
Brief Title: Effects of Inhaled Treprostinil on Exercise Performance in Exercise Induced Pulmonary Hypertension
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Principal Investigator, Timothy Fernandes, Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 813050; ISS-2025-0061 (Other Grant/Funding Number: United Therapeutics)
Record Dates: First submitted 2025-08-07; First posted 2025-08-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Hypertension
Keywords: Exercise Induced Pulmonary Hypertension; Tyvaso; Inhaled treprostinil; Cardiopulmonary exercise testing
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Single arm, every participant will receive inhaled treprostinil
  Interventions: Drug: Inhaled treprostinil

INTERVENTIONS:
Drug: Inhaled treprostinil — Inhaled treprostinil is an inhaled prostacyclin analog which triggers pulmonary arterial dilation. This is the only intervention in this trial.
  Other Names: tyvaso

SUMMARY:
This study aims to investigate therapies for exercise induced pulmonary hypertension (EiPH). This is a condition that effects the blood vessels in the lungs and causes shortness of breath with activity. Currently, there are very limited treatment options for this condition. Inhaled treprostinil, also known as Tyvaso, is a medication used to treat other forms of lung disease and is safe and well tolerated. This study will measure the ability of Tyvaso to improve symptoms related to EiPH and improve performance on exercise testing.

DETAILED DESCRIPTION:
Exercise-induced pulmonary hypertension (EiPH) is defined by the presence of normal resting pulmonary hemodynamics with an abnormal elevation in mean pulmonary artery pressure (mPAP) for a given cardiac output with exercise. EiPH is typically characterized by exertional dyspnea, with the absence of other features of resting pulmonary arterial hypertension (PAH) such as elevated right atrial pressure at rest or lower extremity peripheral edema. Since patients with EiPH have normal resting echocardiograms, the disease is often underdiagnosed. Exercise right-heart catheterization remains the gold standard in diagnosing EiPH.

Aside from subjective markers of clinical improvement with therapy, assessment for physiological improvement is challenging since most measures of PAH severity, including echocardiograms, biomarkers and risk calculators, are normal at baseline in this population with EiPH. The investigators have pioneered the use of non-invasive cardiopulmonary exercise testing (CPET) to assess patients with cardiopulmonary limitations during exercise. Changes in oxygen pulse (O2 pulse) during exercise on CPET have previously been validated as an accurate predictor of stroke volume augmentation, which is an important physiological adaptation to exercise, and may serve as an objective marker of improvement in patients with EiPH.

While the guidelines agree that EiPH is real and under-diagnosed, there is no consensus on the management since these patients have not been included in high-quality clinical trials for PAH treatment. Given the lack of treatment guidelines for EiPH, many providers use PAH-targeted therapy off-label in EiPH. Specifically, generic phosphodiesterase-5 inhibitors are the typical first line agent due to insurance barriers to accessing other therapies. Inhaled treprostinil (Tyvaso DPI) would be an ideal medication for this population. Tyvaso DPI is a convenient, inhaled medication with quick onset. The favorable pharmacokinetic profile raises the potential of this medication for dosing prior to exertion for patients with EiPH.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Persons, aged 18 years of older
* Established diagnosis of exercise induced pulmonary hypertension defined by the following:

  1. Invasive cardiopulmonary exercise testing demonstrating a mean pulmonary artery pressure to cardiac output (P/Q slope) greater than 3 mmHg/L/min
  2. Symptoms of exertional dyspnea
* Ability to perform non-invasive cardiopulmonary exercise testing, either on upright bicycle or treadmill
* If childbearing age, patient must agree to use of effective contraception during the trial

Exclusion Criteria:

* Diagnosis of pulmonary hypertension as defined by resting mean pulmonary arterial pressure of ≥ 20 mmHg, PVR > 3
* Severe underlying chronic lung disease (e.g. COPD, interstitial lung disease)
* Underlying chronic left ventricular disease (e.g. heart failure with reduced ejection fraction)
* Chronic thromboembolic disease
* Pregnancy
* Acute infectious symptoms including fevers within the last week
* Inability or unwillingness to discontinue any phosphodiesterase 5 inhibitors or other off-label
* Known allergic reactions to inhaled treprostinil
* Inability to comply with study protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Stroke volume augmentation before and after inhaled treprostinil | 30 minutes after initial dose of inhaled treprostinil
  Stroke volume augmentation is a physiologic parameter which reflects the hearts ability to respond to physiologic demands of exercise. Stroke volume can be inferred during cardiopulmonary exercise testing by calculating the O2 pulse. Oxygen uptake (VO2) and heart rate are directly measured during cardiopulmonary exercise testing. O2 pulse is calculated by dividing VO2 by heart rate. Stroke volume augmentation is the ratio of O2 pulse at baseline (at the beginning of exercise) and at anaerobic threshold. Stroke volume augmentation will be measured before and after treatment with inhaled treprostinil to assess for improvements in heart function during exercise.

SECONDARY OUTCOMES:
PAH Sympact Scoring | 8 weeks
  PAH Sympact is a validated symptom assessment questionnaire, measuring patient reported outcomes related to cardiopulmonary symptoms and impact on daily life. Each domain is assessed a score from 0-4, with higher numbers representing more severe symptomatology of limitation. This questionnaire will be completed by the participants before initiation of inhaled treprostinil and after 8 weeks of therapy.
Long term stroke volume augmentation | 8 weeks
  Stroke volume augmentation (see description in primary outcomes description) will be retested after 8 weeks of therapy with inhaled treprostinil
Dead space ventilation | 30 minutes, 8 weeks
  Dead space ventilation is a measure of ventilatory efficiency. This is assessed during cardiopulmonary exercise testing through continuous measurement of exhaled carbon dioxide and monitoring of tissue carbon dioxide levels. It will be measured before treatment with inhaled treprostinil, 30 minutes after the first dose of treprostinil, and again after 8 weeks of treprostinil therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Fernandes, MD, Principal Investigator — University of California, San Diego

IPD SHARING:
Plan to Share IPD: Yes
Patients name, phone number, and medical record number will be stored with associated information regarding baseline diagnostic testing, cardiopulmonary exercise testing results, PAH-Sympact scores, and adverse event reporting
Supporting Information: Study Protocol, ICF
Time Frame: IPD and supporting information will be available from trial start date (previously specified) until two years after study completion date (previously specified)
Access Criteria: IPD will be stored on a password protected RedCap database and analyzed on password protected and encrypted devices belonging to the University of California, San Diego or the study team. Only members of the study team will be able to access IPD. Any other dissemination of IPD will be shared in a manner that is de-identified. Publication of individual results may occur but this will be presented in a de-identified manner (ie through individual data points on a spaghetti plot).